CLINICAL TRIAL: NCT04096755
Title: Targeted Metabolic Profiling in Deep Vein Thrombosis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 245270
Record Dates: First submitted 2019-07-15; First posted 2019-09-20 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Deep Vein Thrombosis
Keywords: Deep Vein Thrombosis
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine and serum samples will be obtained from participants for Nuclear Magnetic Resonance Spectroscopy and Mass Spectroscopy analysis. We will retain serum samples from the DVT patients for future DNA research (not part of this project)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DVT group: 40 patients with a confirmed deep venous thrombosis (DVT) on Duplex ultrasound will be recruited into this group. All patients will have serum and urine samples for analysis.
  Interventions: Diagnostic Test: Procedure
- Control Group: 40 volunteers without a DVT will be recruited for the control group. They will have urine and serum samples taken for analysis.
  Interventions: Diagnostic Test: Procedure

INTERVENTIONS:
Diagnostic Test: Procedure — serum and urine samples will be taken for analysis

SUMMARY:
Deep venous thrombosis(DVT) is a blood clot, usually affecting the legs, causing pain, swelling, and redness. The clot damages the veins, which can result in chronic pain, swelling and ulceration. This is called the post-thrombotic syndrome, which impacts heavily on patients' life and work. If the clot dislodges and travels to the lungs, it becomes a pulmonary embolus (PE), which can be life threatening. Together, DVT and PE affect 500,000 people in Europe every year, representing the most common cause of hospital acquired death. They are expensive diseases due to the cost of treatment and the days lost from people being unable to work.

DVT is diagnosed by clinical examination, risk scoring and a blood test called D dimer, a product of the clot. If negative, it is unlikely that DVT is present. However, many conditions can raise D-dimer levels, making it less useful when positive. Ultrasound can confirm the presence of clot but often this is not seen. The clot can take time to form and patients may not experience symptoms immediately. This is a problem for treatment, as new, clot-busting medication works best in the first 2 weeks after a DVT and it is difficult to tell when the clot formed.

Metabonomics is highly sensitive technology that detects very small chemicals; it is being used successfully in cancer and is a tool that can help better understand DVT and generate new tests to help patients.

Previous departmental work has shown that a chemical difference exists in patients with DVT. The aim of this study is to not only confirm the presence of these chemicals in a different group of DVT patients, but also to calculate chemical concentrations. This will improve the investigator's understanding of how DVT develops and provide a way to develop a test that is better than D-dimer.

DETAILED DESCRIPTION:
Deep venous thrombosis (DVT) is a blood clot, usually affecting the legs, causing pain, swelling, and redness. The clot damages the veins, which can result in chronic pain, swelling and ulceration. This is called the post-thrombotic syndrome, which impacts heavily on patients' life and work. If the clot dislodges and travels to the lungs, it becomes a pulmonary embolus (PE), which can be life threatening. Together, DVT and PE affect 500,000 people in Europe every year, representing the most common preventable cause of hospital acquired death. They are expensive conditions not only due to their treatment costs, but also secondary to the resulting loss of work days and productivity.

DVT is diagnosed by clinical examination, risk scoring, usually via the Wells Score, and a blood test called D dimer, a fibrin degradation product. D-dimer is specific but not very sensitive. In other words, when the test is negative, it is unlikely that a DVT is present.

However, many conditions can raise D-dimer levels, making it less useful when positive. Duplex ultrasound can confirm the presence of clot but this can be difficult to visualize or is often not seen at all. The clot can take time to form and patients may not experience symptoms immediately. This is a problem for treatment, as new, clot-busting medication works best in the first 2 weeks after a DVT and it is currently impossible to tell when the thrombus formed.

Because of the importance of DVT, and ongoing issues regarding its diagnosis, ageing and prognosis, numerous research groups have been exploring novel candidate biomarkers to help develop a more accurate diagnostic and prognostic marker for DVT. The Section of Vascular Surgery and of Computational and Systems Medicine (CSM) at Imperial College, have had a longstanding collaboration working towards this end using metabonomics.

Metabonomics is defined as: 'the quantitative measurement of the multiparametric metabolic response of living systems to pathophysiological stimuli or genetic modification'. In other words, it examines the end products of cellular metabolism via platforms such as Nuclear Magnetic Resonance Spectroscopy (NMR) and Mass Spectrometry (MS), which are both high throughput analytical platforms. These enable the qualification (untargeted) and quantification (targeted) of different molecules in a given sample, to a degree of detail superior to that offered by other omic technologies (e.g. proteomics). Metabonomics has demonstrated clear applications in vascular disease, including chronic venous disease , atherosclerosis , venous leg ulceration, aneurysmal disease and stroke.

Untargeted preliminary work on deep venous thrombosis has revealed a metabolic signature for DVT using a murine animal model [9], and promising pilot data in a human study. The aim of the proposed study is to validate previous findings in a separate patient cohort and perform quantification of the metabolites identified in the pilot studies via targeted NMR and MS experiments, continuing the exploration of novel biomarkers for DVT.

Study Design

The study is a prospective observational case-control study, recruiting 40 DVT patients and 40 healthy subjects. Patients diagnosed with a DVT will be recruited at the sites of Imperial College Healthcare NHS Trust.

Summary Forty patients diagnosed with a DVT will be recruited. Participation in the study will not interfere with the decision making and diagnostic investigations by the direct care team. A second control group of 40 healthy volunteers will be also examined. Healthy subject recruitment will take place at the same sites. A patient information leaflet will be provided to participants for informed consent purposes.

A member of the research team will explain the study to prospective participants. Both patients and volunteers will be given sufficient time to read the information sheet and make an informed decision regarding participation in the study; this will be confirmed by the participant signing a consent form. The study involves a comprehensive history and clinical examination, recording medication taken and collection of blood and urine samples. The samples will be labeled anonymously with a study number and transferred to the Imperial

College laboratories in South Kensington. Sample transfer will be performed securely according to established departmental standard operating procedures (SOPs). A blood sample will be stored for future DNA analysis in DVT patients to complement the findings from the metabonomic assays. No DNA analysis will be performed for this particular project.

The DVT group will have a repeat ultrasound study, performed by a vascular research fellow on a dedicated (non-NHS) machine 3 weeks after anticoagulation treatment has ended. They will also have repeat urine and blood samples taken. None of the research interventions will have an impact on the clinical care the patients will receive.

A letter explaining the purpose of the study will be sent to the General Practitioner if the participant wishes. All clinical and research information will remain confidential.

Patient Groups:

* Group 1: Patients with DVT confirmed by lower limb venous duplex ultrasound (DUS) (n =40)
* Group 2: Healthy volunteers with no DVT confirmed on DUS (n = 40)

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* Willing/able to give written informed consent
* Patients with DVT and age and sex matched controls confirmed on duplex ultrasound

Exclusion Criteria:

* Pregnancy (excluded based upon patient history, documented last menstrual period and urinary pregnancy test if patient unsure)
* Patients with blood borne disorders (HIV, Hepatitis B, C)
* Patients on systemic steroids and immunomodulating drugs
* Patients involved in a different venous research project or who have recently been involved with a venous research project

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All study participants will be over the age of 18 and have capacity to consent.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Identification of diagnostic deep vein thrombosis metabolites | 24 months
  We are looking for a unique metabolic signature (a change in the concentration of two or more metabolites) in patients with deep vein thrombosis

SECONDARY OUTCOMES:
To validate previously identified molecules/chemicals that were found to differ in the DVT population in comparison to the non DVT controls | 24 months
To establish the concentration of the identified molecules in DVT patients and controls | 24 months
Correlation of identified metabolite concentrations to known DVT biomarkers (e.g. D dimer) | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Alun Davies, Principal Investigator — Imperial College London
Locations (1):
- Imperial College London, Academic Section of vascular Surgery, 4th floor East Wing, Charing Cross Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-05-14): https://cdn.clinicaltrials.gov/large-docs/55/NCT04096755/Prot_SAP_000.pdf
  • Informed Consent Form (2018-11-11): https://cdn.clinicaltrials.gov/large-docs/55/NCT04096755/ICF_001.pdf